CLINICAL TRIAL: NCT04119882
Title: Early Detection of Myocardial Ischaemia in Suspected Acute Coronary Syndromes by Apo J-Glyc as a Novel Pathologically-based Ischaemia Biomarker
Brief Title: Early Detection of Myocardial Ischaemia in Suspected Acute Coronary Syndromes by Apo J-Glyc
Acronym: EDICA
Status: Completed | Type: Observational
Sponsor: Glycardial Diagnostics S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: EDICA_2019
Record Dates: First submitted 2019-10-01; First posted 2019-10-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Ischemia
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Diagnosis; Prognosis; Risk stratification
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Myocardial Infarction; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for ischaemia: Blood test for 121 patients with confirmed cardiac ischemic event
  Interventions: Diagnostic Test: Blood collection
- Negative for ischaemia: Blood test for 283 patients with no cardiac ischemic event
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Blood collection — New biomarker test

SUMMARY:
The objective of the study is to assess the performance characteristics of Apo J-Glyc as a novel biomarker for the early detection of myocardial ischaemia in patients with suspected acute coronary syndromes.

DETAILED DESCRIPTION:
This in vitro diagnosis clinical validation will test the Performance Characteristics of Apo J-Glyc measured with a novel in vitro diagnostic (IVD) test. Blood samples from eligible consenting subjects will be collected at hospital admission, throughout different post admission times (1h, 3h, 24h and 72h or discharge). The quantification of circulating Apo J-Glyc levels will be analysed in correlation with clinical data providing information about Apo J-Glyc as an ischaemia biomarker and its diagnostic and 6-months prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 18 years old
* Chest pain of suspected cardiac origin
* Signature of informed consent
* Able and willing to comply with study requirements

Exclusion Criteria:

* Prior inclusion in the same study
* Life expectancy less than 6 months
* Previous inclusion in a therapy-related clinical trial (except clinical trials testing Medical Devices such as stents and/or balloons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to the Emergency Department (ED) with chest pain of suspected cardiac origin
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia | 0 hour
  Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia as compared to final diagnosis at discharge following routine practice to manage chest pain patients with possible ACS.
Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia | 1 hour
  Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia as compared to final diagnosis at discharge following routine practice to manage chest pain patients with possible ACS.
Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia | 3 hours
  Cut-off value point of Apo J-Gly levels at admission for the early diagnosis of cardiac ischaemia as compared to final diagnosis at discharge following routine practice to manage chest pain patients with possible ACS.
Area under the Receiver Operating characteristic Curve (A-ROC curve) | 0 hour
  Area under the Receiver Operating characteristic Curve will be used to determine the optimum clinical sensitivity and specificity. Results will be generated from subject's blood collected at different collection time points.
Area under the Receiver Operating characteristic Curve (A-ROC curve) | 1 hour
  Area under the Receiver Operating characteristic Curve will be used to determine the optimum clinical sensitivity and specificity. Results will be generated from subject's blood collected at different collection time points.
Area under the Receiver Operating characteristic Curve (A-ROC curve) | 3 hours
  Area under the Receiver Operating characteristic Curve will be used to determine the optimum clinical sensitivity and specificity. Results will be generated from subject's blood collected at different collection time points.
Sensitivity | 0 hours
  Sensitivity results will be generated from subject's blood collected at different collection time points.
Sensitivity | 1 hours
  Sensitivity results will be generated from subject's blood collected at different collection time points.
Sensitivity | 3 hours
  Sensitivity results will be generated from subject's blood collected at different collection time points.
Specificity | 0 hour
  Specificity results will be generated from subject's blood collected at different collection time points.
Specificity | 1 hour
  Specificity results will be generated from subject's blood collected at different collection time points.
Specificity | 3 hours
  Specificity results will be generated from subject's blood collected at different collection time points.
Negative Predictive Value (NPV) | 0 hour
  Negative Predictive Value results will be generated from subject's blood collected at different collection time points.
Negative Predictive Value (NPV) | 1 hour
  Negative Predictive Value results will be generated from subject's blood collected at different collection time points.
Negative Predictive Value (NPV) | 3 hour
  Negative Predictive Value results will be generated from subject's blood collected at different collection time points.
Positive Predictive Value (PPV) | 0 hour
  Positive Predictive Value results will be generated from subject's blood collected at different collection time points.
Positive Predictive Value (PPV) | 1 hour
  Positive Predictive Value results will be generated from subject's blood collected at different collection time points.
Positive Predictive Value (PPV) | 3 hours
  Positive Predictive Value results will be generated from subject's blood collected at different collection time points.

SECONDARY OUTCOMES:
Prognosis and risk-stratification. Incidence of Major following Adverse Cardiac Event (MACE). | From admission to up to 6 months
  Subjects will be assessed for the in-hospital and 6-month incidence of any Major following Adverse Cardiac Event (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Judit Cubedo, Study Director — Glycardial Diagnostics
Locations (10):
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Álvaro Cunqueiro de Vigo, Vigo
- United Kingdom (2):
  - Chelsea and Westminister Hospital NHS Foundation Trust, London
  - East & North Hertfordshire NHS Trust, Lister Hospital, Stevenage